CLINICAL TRIAL: NCT00120913
Title: Continuous Oral Contraceptives (COCs): Are Bleeding Patterns Dependent on the Hormones Given?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: OHSU IRB 7198
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2005-07-19 (Estimated); Status verified 2005-07

CONDITIONS: Breakthrough Bleeding
Keywords: Breakthrough bleeding while taking continuously dosed oral contraceptives
MeSH Terms: conditions — Metrorrhagia | interventions — Contraceptives, Oral

INTERVENTIONS:
Drug: Birth control pills

SUMMARY:
While there may be a decrease in the total number of bleeding days women experience with continuous-dosed COCs (no menstrual withdrawal week), these regimens frequently result in an increased number of "breakthrough" or non-scheduled bleeding days. Breakthrough bleeding is among the main reasons cited for discontinuation of combined COCs dosed traditionally (3 weeks of active pill, 1 week of placebo) or continuously, and may offset the perceived benefit of fewer withdrawal bleeding events for many women taking continuous-dosed COCs. The exact mechanisms responsible for breakthrough bleeding patterns during hormonal contraception are unknown and may be related to the pill formulation. This study is to determine whether progestin type or estrogen dose influences bleeding patterns, side effects, or satisfaction with combined oral contraceptives (COC) dosed continuously.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 to 49 years old
* Good general health
* No medical contraindications to combined COC therapy.
* In addition, all participants were required to have taken cyclic COCs for at least three months at the time of enrollment, in order to avoid common transition bleeding with the initiation of COCs.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160
Dates: Study Completion 2004-08

PRIMARY OUTCOMES:
Bleeding patterns

SECONDARY OUTCOMES:
Satisfaction, menstrual-associated symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Alison B Edelman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States